CLINICAL TRIAL: NCT00906724
Title: An Exercise Intervention in Insulin-Resistant Minority Adolescents
Brief Title: An Exercise Intervention Study in Insulin-Resistant Adolescents
Acronym: 3290
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Eric Paul Hoffman, Children's National Medical Center
Other Study IDs: U10HD030447 (NIH)
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-01

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Exercise; insulin resistance factor (uremia); Adiposity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aerobic exercise: Aerobic exercise in Insulin Resistant Minority Adolescents
  Interventions: Procedure: Aerobic exercise

INTERVENTIONS:
Procedure: Aerobic exercise — A graded exercise stress test (GXT) will be done under cardiologist supervision.
  Subjects will undergo three month of supervised aerobic exercise.
  Other Names: Insulin Resistance; Obesity; Exercise

SUMMARY:
Hypothesis: Insulin-resistant African-American and Hispanic adolescents will show significant improvement of insulin sensitivity (SI) and positive changes associated with fibrinolytic markers and lipid profile after a two month supervised aerobic training.

DETAILED DESCRIPTION:
The specific aims of the study are 1) To determine the effects of exercise on insulin sensitivity in insulin-resistant African-American and Hispanic adolescents; 2) To determine the effects of exercise on fibrinolytic markers in insulin-resistant African-American and Hispanic adolescents.

The hypothesis is that insulin-resistant African-American and Hispanic adolescents will show significant improvement of insulin sensitivity (SI) and positive changes associated with fibrinolytic markers and lipid profile after a 1 month pre-training period and two-months of supervised, moderate intensity aerobic exercise.

Part I. Insulin-resistant African American and Hispanic adolescents from the DC metro area will be recruited through various recruitment efforts. Potential participants will have 2 screening visits in which their medical history, physical activity level, body mass index, and fasting plasma glucose and insulin or OGTT results will determine eligibility.

Part 2. If inclusion criteria is met, the subjects will undergo a 2 week dietary stabilization period, treadmill exercise testing, IVGTT, blood draws for fibrinolytic and lipid markers, DEXA scan, and anthropometric measurements. Subjects will have a 1 month pre-training period and 2 months of supervised, moderate intensity aerobic exercise. All baseline testing will be repeated after the exercise period to see any significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 14 to 18 years old
* Being African American or Hispanic
* Sedentary (exercising less than twice a week for less than 20 minutes)
* Non-smoker
* At high risk of developing insulin resistance
* BMI for age grater than or equal to the 95th percentile

Exclusion Criteria:

* History of chronic illnesses
* Thyroid dysfunction
* Taking medications know to affect metabolism
* Being pregnant or lactating

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Insulin-Resistant Minority Adolescents
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity index | 6 month

SECONDARY OUTCOMES:
Levels of change in fibrinolytic markers | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Hoffman, PHD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States